CLINICAL TRIAL: NCT01476631
Title: Step Down Colon Cancer Risk: A Pilot Intervention for Colon Cancer Risk Reduction
Brief Title: Step Down Colon Cancer Risk
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough patients consented during the funding period
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201105308
Record Dates: First submitted 2011-11-09; First posted 2011-11-22 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Adenomatous Polyps
MeSH Terms: conditions — Adenomatous Polyps | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: 30 minutes walking (Experimental): First Step program with 30 minutes of walking and 10,000 steps per day for 3 months.
  Interventions: Behavioral: Walking
- Arm B: 60 minutes walking (Experimental): First Step program with 60 minutes of walking and 13,000 steps per day for 3 months.
  Interventions: Behavioral: Walking

INTERVENTIONS:
Behavioral: Walking — * 7 days prior to baseline participants must wear a blinded pedometer
  * At baseline information on the blinded pedometer will downloaded to the computer for analysis as well as number of days worn and hours of wear. Sociodemographic, cancer risk factors, height/weight, fast blood draw to check levels on insulin, C-peptide, IL-6 and PEG-2 and questionnaires PPAQ, Exercise Confident Survey and Sallis Social Support Scale, Day/night; Home/Work, neighborhood safety, HINTS, IPAPS, CES-D, Brief COPE, Urban and Life Stress Scale.

SUMMARY:
Hypothesis 1: Exercise will decrease serum markers in a dose response manner.

Hypothesis 2: Participants in the 60 minute intervention will have significantly higher physical activity levels than those in the 30 minute intervention at three months.

DETAILED DESCRIPTION:
Primary Aim: To conduct a dose response pilot trial of low (30 min/day) or high (60 min/day) dose exercise in men and women at increased risk of colon cancer. The major outcomes are changes in serum levels of four risk-related biomarkers: insulin, C-peptide, IL-6 and PGE-2.

Secondary Aim. To compare changes in the secondary outcome of physical activity over three months.

ELIGIBILITY:
Inclusion Criteria:

* aged 50 to 80
* no personal cancer history
* found to have an adenomatous polyp upon colonoscopy at BJH/WUSM in the previous six months
* no contraindications to beginning an exercise program
* no previous diagnosis of familial polyposis syndromes
* no previous diagnosis of ulcerative colitis or Crohn's disease;

Exclusion Criteria:

* Participants who are regular NSAID users will be excluded as this may interfere with the measurement of inflammatory marker outcomes. Regular use is defined as taking 80mg or more per day of aspirin, ibuprofen, naproxen or other NSAID 5 or more days of the week.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Exercise will decrease serum markers (insulin, C-peptide, IL-6 and PGE-2) in a dose response manner. | 3 months
  Changes in serum levels of four risk-related biomarkers: insulin, C-peptide, IL-6 and PGE-2 comparing baseline and 3 months serum levels.

SECONDARY OUTCOMES:
Participants in the 60 minute intervention will have significantly higher physical activity levels (measured by pedometer and accelerometer) than those in the 30 minute intervention at three months. | 3 months
  Comparing changes in the secondary outcome of physical activity over three months, as measured by pedometer and accelerometer.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Y. Wolin, ScD, FACSM, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Wolin KY, Fagin C, James AS, Early DS. Promoting physical activity in patients with colon adenomas: a randomized pilot intervention trial. PLoS One. 2012;7(7):e39719. doi: 10.1371/journal.pone.0039719. Epub 2012 Jul 13. PMID 22808053
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu